CLINICAL TRIAL: NCT06340815
Title: Varian ProBeam Proton Therapy System Clinical Trial (Shandong)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2022-02
Record Dates: First submitted 2024-03-22; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Tumor, Solid
Keywords: Tumor; Radiation therapy; Proton therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: a clinical study of prospective, single-arm objective performance criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm objective performance criteria (OPC) (Experimental): According to the NMPA Guidance on Proton and Carbon Ion treatment system clinical evaluation and clinical trial, the objective performance criteria for the validity of medical device treatment for trial use should be at least 80%, with an expected target of 95% in which the validity is defined as: Complete Response (CR) + Partial Response (PR)+ Stable Disease (SD), and the definition of tumor disease control rate in this clinical trial is basically identical. Therefore, the clinical trial did not have a control group, but using single-arm objective performance criteria, when evaluating ProBeam radiotherapy for tumor patients, the main validity evaluation index of tumor disease control rate; the main safety evaluation by incident of acute radiation injury and adverse event.
  Interventions: Device: Radiation: Proton Therapy System (ProBeam)

INTERVENTIONS:
Device: Radiation: Proton Therapy System (ProBeam) — All enrolled subjects will be treated with Proton radiation therapy using the medical device Varian Proton Therapy System (ProBeam). The screening period from informed consent to enrollment is expected to be 2 weeks, while the treatment period depends on patient medical situation and treatment plan. The period after the last treatment is divided into short-term follow-up which is 90 days after treatment completion and long-term follow-up which is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for NMPA regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up is finished.
  And long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.

SUMMARY:
This study is prospective, single-center, single-arm objective performance criteria.

This trial will be conducted with a total of 47 subjects enrolled. All of subjects will be treated with radiation therapy using the medical device Varian ProBeam Proton Therapy System (ProBeam), aim to compare the data with objective performance criteria (OPC) to evaluate the effectiveness and safety of ProBeam radiotherapy system for oncology patients, providing a clinical basis for the medical device registration.

DETAILED DESCRIPTION:
Oncology patients, including tumors of head and neck, chest, abdomen, spine, pelvic cavity, extremities and other tumors. The screening period from informed consent to enrollment is expected to be 2 weeks, while the treatment period depends on patient medical situation and treatment plan. The period after the last treatment is divided into short-term follow-up which is 90 days after treatment completion and long-term follow-up which is 5 years after treatment completion. The clinical trial with short-term follow-up fulfills the requirements for National Medical Products Administration (NMPA) regulatory registration. All the end points claimed will be achieved in the short-term follow-up stage. The trial is defined as completion once short-term follow-up is finished.

And long-term follow-up report will be submitted for future post market evaluation when requested by NMPA.

ELIGIBILITY:
Inclusion Criteria (Major Criteria):

1. Patients diagnosed with histological/pathological diagnosis and/or with imaging, laboratory examination and other evidence, clinically diagnosed as benign and malignant intracranial tumors, and malignant solid tumors of the head and neck, chest, abdomen, spine, pelvis, and extremities;
2. Eastern Cooperative Oncology Group (ECOG) physical condition grade ≤ 2;
3. Women of childbearing had negative results in the blood pregnancy test (Human Chorionic Gonadotropin, HCG) 7 days prior to the first treatment;
4. The subject or subject's guardian is able to understand the purpose of the study, demonstrate sufficient compliance with the protocol and sign informed consent form.

Exclusion Criteria (Major Criteria):

1. There are contraindications to radiation therapy, including congenital susceptibility to ionizing radiation hypersensitivity; or the presence of comorbidity that may lead to ionizing radiation hypersensitivity, which will increase the sensitivity of normal tissues to radiation therapy;
2. The tumor recurring at the same site has received two or more radiotherapy treatments;
3. Active implants such as cardiac pacemakers, defibrillators, cochlear implants, drug infusion pumps, other nerve stimulators, etc. (whether they are turned on or not) within the scope of radiotherapy ; or passive implants that affect radiotherapy thing;
4. Other situations that investigator determines not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness evaluation: Local tumor control rate at 90 days after the proton radiation treatment completion | 90 days ± 7 days after treatment completion
  At 90 days after the end of treatment, the number of cases in partial response (PR) and stable disease (SD) and complete response (CR) accounted for the proportion of total cases will be graded based on Response Evaluation Criteria in Solid Tumors RECIST Version 1.1 (RECIST 1.1) criteria.
Safety evaluation: Incidence of Acute radiation injury | from enrollment to 90 days ± 7 days after treatment completion
  Observe acute radiation injury occurrence throughout the trial period, including the treatment period and the 90-day follow-up period. Acute radiation injury will be summarized separately (calculating quantity of participants, number of cases, and incidence) based on Radiation Therapy Oncology Group (RTOG) Grading Criteria.
Safety evaluation: Incidence of Adverse Events based on CTCAE 5.0 criteria | from enrollment to 90 days ± 7 days after treatment completion
  record Incidence of Adverse Events and estimate according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0) criteria, level 3 toxic reaction ratio should be lower than the acceptable value (5%), level 4 and 5 toxic reaction should not occur.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Sophia Shao, Shanghai, China

IPD SHARING:
Plan to Share IPD: No